CLINICAL TRIAL: NCT02584504
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Alirocumab in Patients With Hypercholesterolemia Not Adequately Controlled With Non-statin Lipid Modifying Therapy or the Lowest Strength of Statin
Brief Title: Efficacy and Safety of Alirocumab in Patients With Hypercholesterolemia Not Adequately Controlled With Non-statin Lipid Modifying Therapy or the Lowest Strength of Statin
Acronym: ODYSSEY-NIPPON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14305; U1111-1170-7697 (Other: UTN)
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Hypercholesterolemia
Keywords: Non-statin LMT; Low dose statin
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Atorvastatin; Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Alirocumab 150 mg Q4W (Experimental): Double-blind treatment period(DBTP):participants received Alirocumab 150 mg subcutaneous injection every 4 week(Q4W) alternating with placebo(for alirocumab)Q4W added to lowest-strength statin therapy(atorvastatin 5 mg daily),stable non-statin LMT/diet therapy alone for 12weeks. Participants completed DBTP,entered open-label treatment period(OLTP),received alirocumab 150 mg Q4W up to additional 52 weeks. Alirocumab dose up-titrated to 150 mg every 2 weeks(Q2W) at Week 24(OLTP:Week 12),when targeted LDL-C level at Week 20 not achieved as Japan Atherosclerosis Society Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012:1) ≥100 mg/dL(2.59 mmol/L) in heterozygous familial hypercholesterolemia (heFH) participants/non-familial hypercholesterolemia (non-FH)participants with history of documented coronary heart disease;2) ≥120 mg/dL(3.10 mmol/L)in non-FH participants with history of documented diseases/other risk factors as categorized in primary prevention category III)
  Interventions: Drug: Alirocumab; Drug: Placebo; Drug: Atorvastatin; Drug: Non-statin Lipid-Modifying Therapy; Other: Diet Alone
- Alirocumab 150 mg Q2W (Experimental): In DBTP, participants received Alirocumab 150 mg subcutaneous (SC) injection Q2W added to lowest-strength statin therapy (atorvastatin 5 mg daily), stable non-statin LMT or diet therapy alone for 12 weeks. Participants who completed DBTP were entered in OLTP and received alirocumab 150 mg Q4W up to additional 52 weeks. Alirocumab dose up-titrated to 150 mg Q2W at Week 24 (Week 12 of OLTP), when targeted LDL-C levels at Week 20 were not achieved i.e. LDL-C ≥100 mg/dL (2.59 mmol/L) or ≥120 mg/dL (3.10 mmol/L) according to Japan Atherosclerosis Society(JAS) Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin; Drug: Non-statin Lipid-Modifying Therapy; Other: Diet Alone
- Placebo Q2W (Placebo Comparator): In DBTP, participants received Placebo (for alirocumab) SC injection Q2W added to lowest-strength statin therapy (atorvastatin 5 mg), stable non-statin LMT or diet therapy alone for 12 weeks. Participants who completed DBTP were entered in OLTP and received alirocumab 150 mg Q4W up to additional 52 weeks. Alirocumab dose up-titrated to 150 mg Q2W at Week 24 (Week 12 of OLTP), when targeted LDL-C levels at Week 20 were not achieved i.e. LDL-C ≥100 mg/dL (2.59 mmol/L) or ≥120 mg/dL (3.10 mmol/L) according to JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
  Interventions: Drug: Placebo; Drug: Atorvastatin; Drug: Non-statin Lipid-Modifying Therapy; Other: Diet Alone

INTERVENTIONS:
Drug: Alirocumab — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a disposable auto-injector.
  Other Names: SAR236553; REGN727
  Arms: Alirocumab 150 mg Q2W; Alirocumab 150 mg Q4W
Drug: Placebo — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a disposable auto-injector.
  Arms: Alirocumab 150 mg Q4W; Placebo Q2W
Drug: Atorvastatin — Atorvastatin 5 mg tablet orally.
Drug: Non-statin Lipid-Modifying Therapy — Ezetimibe, Bezafibrate or Fenofibrate at stable dose as background therapy.
Other: Diet Alone — Stable cholesterol-lowering diet as background therapy.

SUMMARY:
Primary Objective:

To demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) by alirocumab administration as add-on therapy to non-statin lipid modifying therapy (LMT) including diet therapy alone or the lowest strength of statin in comparison with placebo after 12 weeks of treatment in participants with hypercholesterolemia.

Secondary Objective:

* To evaluate the effect of two treatment regimens of alirocumab on other lipid parameters: apolipoprotein B (Apo-B), non-high-density lipoprotein cholesterol (non HDL-C), total cholesterol (TC), lipoprotein (a) (Lp[a]), high-density lipoprotein cholesterol (HDL-C), triglyceride (TG), and apolipoprotein A-1 (Apo A-1).
* To evaluate the safety and tolerability of alirocumab administration.
* To evaluate the development of anti-alirocumab antibodies.
* To evaluate the pharmacokinetic and pharmacodynamic profiles of alirocumab administration.
* To evaluate the long-term safety in participants receiving open-label alirocumab administration.

DETAILED DESCRIPTION:
The duration of study per participant was approximately 71 weeks consisting of a run-in period (4 weeks), a screening period (3 weeks), a double-blind treatment period (12 weeks), and an open-label treatment period (52 weeks).

ELIGIBILITY:
Inclusion criteria :

Participants with hypercholesterolemia (heFH or non-FH) receiving non statin LMTs or the lowest strength of statin.

Exclusion criteria:

* LDL-C <100 mg/dL (<2.59 mmol/L) at the screening visit (Week -3) in participants with heFH or in participants with non-FH who have a history of documented coronary heart disease.
* LDL-C <120 mg/dL (<3.10 mmol/L) at the screening visit (Week -3) in participants with non-FH participants who had a history of documented diseases or other risk factors classified as primary prevention category III as defined in JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
* Not on a stable dose of LMT (including diet therapy alone) in the run-in period or the screening period.
* Fasting serum TGs >400 mg/dL (>4.52 mmol/L) at the screening period.
* Systolic blood pressure (BP) >160 mmHg or diastolic BP >100 mmHg at the run-in visit (Week -7) or the screening visit (Week -3) or the randomization visit (Week 0).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (30):
- Japan (30):
  - Investigational Site Number 392028, Ageo-Shi
  - Investigational Site Number 392007, Chūōku
  - Investigational Site Number 392029, Chūōku
  - Investigational Site Number 392014, Fukui-shi
  - Investigational Site Number 392023, Hachioji-Shi
  - Investigational Site Number 392013, Itoshima-Shi
  - Investigational Site Number 392010, Kanazawa
  - Investigational Site Number 392024, Kasuga-Shi
  - Investigational Site Number 392004, Kawanishi-Shi
  - Investigational Site Number 392015, Kitakyushu-Shi
  - Investigational Site Number 392005, Komatsu-Shi
  - Investigational Site Number 392032, Matsudo-Shi
  - Investigational Site Number 392017, Matsumoto-Shi
  - Investigational Site Number 392003, Mito
  - Investigational Site Number 392018, Morioka
  - Investigational Site Number 392009, Moriya-Shi
  - Investigational Site Number 392006, Nagoya
  - Investigational Site Number 392011, Nagoya
  - Investigational Site Number 392019, Nagoya
  - Investigational Site Number 392025, Nagoya
  - Investigational Site Number 392027, Osaka
  - Investigational Site Number 392030, Sakura-Shi
  - Investigational Site Number 392016, Shinagawa-Ku
  - Investigational Site Number 392001, Shinjuku-Ku
  - Investigational Site Number 392008, Shinjuku-Ku
  - Investigational Site Number 392012, Shizuoka
  - Investigational Site Number 392002, Suita-Shi
  - Investigational Site Number 392031, Suita-Shi
  - Investigational Site Number 392020, Toyonaka-Shi
  - Investigational Site Number 392022, Yakushi

REFERENCES:
- [Background] Teramoto T, Kondo A, Kiyosue A, Harada-Shiba M, Ishigaki Y, Tobita K, Kawabata Y, Ozaki A, Baccara-Dinet MT, Sata M. Efficacy and safety of alirocumab in patients with hypercholesterolemia not adequately controlled with non-statin lipid-lowering therapy or the lowest strength of statin: ODYSSEY NIPPON study design and rationale. Lipids Health Dis. 2017 Jun 17;16(1):121. doi: 10.1186/s12944-017-0513-7. PMID 28623954
- [Derived] Teramoto T, Kiyosue A, Ishigaki Y, Harada-Shiba M, Kawabata Y, Ozaki A, Baccara-Dinet MT, Sata M. Efficacy and safety of alirocumab 150mg every 4 weeks in hypercholesterolemic patients on non-statin lipid-lowering therapy or lowest strength dose of statin: ODYSSEY NIPPON. J Cardiol. 2019 Mar;73(3):218-227. doi: 10.1016/j.jjcc.2018.10.004. Epub 2018 Nov 30. PMID 30509509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 30 active centers in Japan. Overall 241 participants were screened between 30 November 2015 and 19 October 2016, of whom 78 were screen failures and 163 were randomized. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization stratified per background statin therapy (Yes/No). "No statin" also stratified per background fibrate/ezetimibe therapy (Yes/No), 'Yes' =fibrate/ezetimibe, 'No' =diet therapy alone. Randomization followed 1:1:1 ratio (Alirocumab 150 mg Q4W: Alirocumab 150 mg Q2W: Placebo Q2W).
Groups:
- Alirocumab 150 mg Q4W: In double-blind treatment period (DBTP), participants received Alirocumab 150 mg subcutaneous (SC) injection every 4 weeks (Q4W) alternating with placebo (for alirocumab) Q4W added to lowest-strength statin therapy (atorvastatin 5 mg daily), stable non-statin Lipid-Modifying Therapy (LMT) or diet therapy alone for 12 weeks. Participants who completed DBTP, entered in open-label treatment period (OLTP) and received alirocumab 150 mg Q4W up to additional 52 weeks (up to Week 64). Alirocumab dose up-titrated to 150 mg every 2 weeks (Q2W) at Week 24 (Week 12 of OLTP), when LDL-C levels ≥100 mg/dL (2.59 mmol/L) or ≥120 mg/dL (3.10 mmol/L) at Week 20 according to Japan Atherosclerosis Society (JAS) Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
- Alirocumab 150 mg Q2W: In DBTP, participants received Alirocumab 150 mg SC injection Q2W added to lowest-strength statin therapy (atorvastatin 5 mg), stable non-statin LMT or diet therapy alone for 12 weeks. Participants who completed DBTP were entered in OLTP and received alirocumab 150 mg Q4W up to additional 52 weeks (up to Week 64). Alirocumab dose up-titrated to 150 mg Q2W at Week 24 (Week 12 of OLTP), when LDL-C levels ≥100 mg/dL (2.59 mmol/L) or ≥120 mg/dL (3.10 mmol/L) at Week 20 according to JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
- Placebo Q2W: In DBTP, participants received Placebo (for alirocumab) SC injection Q2W added to lowest-strength statin therapy (atorvastatin 5 mg), stable non-statin LMT or diet therapy alone for 12 weeks. Participants who completed DBTP were entered in OLTP and received alirocumab 150 mg Q4W up to additional 52 weeks (up to Week 64). Alirocumab dose up-titrated to 150 mg Q2W at Week 24 (Week 12 of OLTP), when LDL-C levels ≥100 mg/dL (2.59 mmol/L) or ≥120 mg/dL (3.10 mmol/L) at Week 20 according to JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
Period: Double-blind Treatment
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Started | 54 (Randomized) | 53 (Randomized) | 56 (Randomized)
ITT Population | 54 | 53 | 56
mITT Population | 54 | 53 | 56
Safety Population | 54 | 53 | 56
Completed | 54 | 51 | 55
Not Completed | 0 | 2 | 1
Not completed — Participant withdrew consent | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Family Matter | 0 | 1 | 0
Period: Open-label Treatment
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Started | 54 | 51 | 55
Treated | 54 | 50 | 54
Completed | 52 | 47 | 47
Not Completed | 2 | 4 | 8
Not completed — Participant withdrew consent | 0 | 0 | 4
Not completed — Adverse Event | 2 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Entered but not treated | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Alirocumab 150 mg Q4W: In DBTP, participants received Alirocumab 150 mg SC injection Q4W alternating with placebo (for alirocumab) Q4W added to lowest-strength of statin therapy (atorvastatin 5 mg daily), stable non-statin LMT or diet therapy alone for 12 weeks. Participants who completed DBTP were entered in OLTP and received alirocumab 150 mg Q4W up to additional 52 weeks (up to Week 64). Alirocumab dose up-titrated to 150 mg Q2W at Week 24 (Week 12 of OLTP), when LDL-C levels ≥100 mg/dL (2.59 mmol/L) or ≥120 mg/dL (3.10 mmol/L) at Week 20 according to Japan Atherosclerosis Society (JAS) Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
- Total: Total of all reporting groups
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W | Total
Number analyzed (Participants) | 54 | 53 | 56 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.8) | 63.6 (10.4) | 64.6 (10.0) | 63.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 19 | 60
  Male | 33 | 33 | 37 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 54 | 53 | 56 | 163
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C in mg/dL from Friedewald formula (LDL cholesterol = Total cholesterol - high density lipoprotein [HDL] cholesterol - [Triglyceride/5]).
  mg/dL | 154.2 (59.5) | 149.2 (31.1) | 149.4 (32.6) | 150.9 (42.8)
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 3.993 (1.541) | 3.865 (0.806) | 3.870 (0.844) | 3.909 (1.109)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12- Intent to Treat (ITT) Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Week 12 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 12 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 12
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Alirocumab 150 mg Q4W: Participants received Alirocumab 150 mg SC injection Q4W alternating with placebo (for alirocumab) Q4W added to lowest-strength of statin therapy (atorvastatin 5 mg daily), stable non-statin LMT or diet therapy alone for 12 weeks in DBTP.
- Alirocumab 150 mg Q2W: Participants received Alirocumab 150 mg SC injection Q2W added to lowest-strength statin therapy (atorvastatin 5 mg), stable non-statin LMT or diet therapy alone for 12 weeks in DBTP.
- Placebo Q2W: Participants received Placebo (for alirocumab) SC injection Q2W added to lowest-strength statin therapy (atorvastatin 5 mg), stable non-statin LMT or diet therapy alone for 12 weeks in DBTP.
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -43.8 (2.2) | -70.1 (2.3) | -4.3 (2.2)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; Alirocumab 150 mg Q4W group was compared to placebo group using an appropriate contrast statement; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; Threshold for significance at 0.025 level; Least Square (LS) Mean Difference = -39.5, 97.5% CI 2-sided [-46.5 to -32.4] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; Alirocumab 150 mg Q2W group was compared to placebo group using an appropriate contrast statement; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -65.8, 97.5% CI 2-sided [-72.9 to -58.7] — Alirocumab 150 mg Q2W vs. Placebo
Statistical Analysis 3: Comparison: Alirocumab 150 mg Q4W vs Alirocumab 150 mg Q2W; Alirocumab 150 mg Q4W group was compared to Alirocumab 150 mg Q2W group using an appropriate contrast statement; Test type: Other — Statistical test was not planned because this comparison was for a descriptive purpose; LS Mean Difference = -26.3, 95% CI 2-sided [-32.5 to -20.0] — Alirocumab 150 mg Q4W group vs Alirocumab 150 mg Q2W

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12- On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 12 (i.e. up to 21 days after last double-blind injection).
Time Frame: From Baseline to Week 12
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -43.4 (2.1) | -70.1 (2.2) | -2.8 (2.1)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.025 level. Hierarchical procedure for comparisons of Alirocumab 150 mg Q4W versus Placebo Q2W and Alirocumab 150 mg Q2W versus Placebo Q2W were processed separately; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -40.6, 97.5% CI 2-sided [-47.4 to -33.8] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant for the relevant compared arms); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -67.4, 97.5% CI 2-sided [-74.2 to -60.5] — Alirocumab 150 mg Q2W vs. Placebo

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C to Averaged Week 10 to 12: ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 12 regardless of status on- or off-treatment and assigning a weight of 0.5 for Week 10 and 12 time points.
Time Frame: From Baseline to Week 12
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -54.2 (1.9) | -69.9 (1.9) | -3.7 (1.9)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -50.5, 97.5% CI 2-sided [-56.6 to -44.5] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -66.2, 97.5% CI 2-sided [-72.3 to -60.1] — Alirocumab 150 mg Q2W vs. Placebo

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C to Averaged Week 10 to 12- On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 12 (i.e. up to 21 days after last double-blind injection) and assigning a weight of 0.5 for Week 10 and 12 time points.
Time Frame: From Baseline to Week 12
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -54.0 (1.9) | -69.9 (1.9) | -2.6 (1.9)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -51.4, 97.5% CI 2-sided [-57.4 to -45.4] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -67.3, 97.5% CI 2-sided [-73.3 to -61.3] — Alirocumab 150 mg Q2W vs. Placebo

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo-B) at Week 12: ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 12 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 12
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -32.2 (2.0) | -57.9 (2.0) | -6.0 (2.0)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -26.2, 97.5% CI 2-sided [-32.5 to -19.9] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -51.9, 97.5% CI 2-sided [-58.3 to -45.5] — Alirocumab 150 mg Q2W vs. Placebo

6. Secondary Outcome: Percent Change From Baseline in Apo-B at Week 12- On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including available post-baseline on-treatment data at from Week 4 to Week 12 (i.e. up to 21 days after last double-blind injection).
Time Frame: From Baseline to Week 12
Population: Participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment (Apo-B mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 55
percent change | -31.8 (2.0) | -58.0 (2.0) | -4.6 (1.9)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -27.2, 97.5% CI 2-sided [-33.5 to -20.9] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -53.4, 97.5% CI 2-sided [-59.7 to -47.1] — Alirocumab 150 mg Q2W vs. Placebo

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12: ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 12
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -36.2 (2.0) | -61.1 (2.0) | -4.9 (2.0)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -31.3, 97.5% CI 2-sided [-37.7 to -25.0] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -56.2, 97.5% CI 2-sided [-62.5 to -49.8] — Alirocumab 150 mg Q2W vs. Placebo

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12- On-treatment Analysis
Description: as for outcome 2
Time Frame: From Baseline to Week 12
Population: Participants of the mITT population with one baseline and at least one post-baseline non-HDL-C value on- treatment (non-HDL-C mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -35.9 (1.9) | -61.1 (2.0) | -3.5 (1.9)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -32.4, 97.5% CI 2-sided [-38.6 to -26.3] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -57.6, 97.5% CI 2-sided [-63.8 to -51.4] — Alirocumab 150 mg Q2W vs. Placebo

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 12- ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 12
Population: Participants of the ITT population with one baseline and at least one post-baseline total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -25.8 (1.5) | -44.7 (1.6) | -3.3 (1.5)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -22.5, 97.5% CI 2-sided [-27.4 to -17.6] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = -41.4, 97.5% CI 2-sided [-46.4 to -36.5] — Alirocumab 150 mg Q2W vs. Placebo

10. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C Goal at Week 12- ITT Analysis
Description: Calculated LDL-C goal was defined as calculated LDL-C <100 mg/dL (2.59 mmol/L) for heterozygous familiar hypercholesterolemia (heFH) participants or non-familial hypercholesterolemia (non-FH) participants who had a history of documented CHD, or <120 mg/dL (3.10 mmol/L) for non-FH participants who had a history of documented diseases or other risk factors as defined in JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012. Adjusted percentages at Week 12 were obtained from multiple imputation approach for handling of missing data. All available post-baseline data from Week 4 to Week 12 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: Up to Week 12
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percentage of participants | 85.2 | 96.2 | 14.3
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.025 level for Bonferroni adjustment; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 61.2, 97.5% CI 2-sided [13.9 to 268.9] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.025 level for Bonferroni adjustment; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 281.4, 97.5% CI 2-sided [33.3 to 2382.2] — Alirocumab 150 mg Q2W vs. Placebo

11. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C Goal at Week 12- On-Treatment Analysis
Description: Calculated LDL-C goal was defined as calculated LDL-C <100 mg/dL (2.59 mmol/L) for heFH participants or non-FH participants who had a history of documented CHD, or <120 mg/dL (3.10 mmol/L) for non-FH participants who had a history of documented diseases or other risk factors as defined in JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012. Adjusted percentages at Week 12 from multiple imputation approach including available post-baseline on-treatment data from Week 4 to Week 12 (i.e. up to 21 days after last double-blind injection).
Time Frame: Up to Week 12
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percentage of participants | 85.2 | 96.2 | 10.8
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.025 level for Bonferroni adjustment; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 102.8, 97.5% CI 2-sided [19.0 to 556.8] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.025 level for Bonferroni adjustment; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 500.8, 97.5% CI 2-sided [47.9 to 5230.9] — Alirocumab 150 mg Q2W vs. Placebo

12. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12: ITT Analysis
Description: Adjusted means and standard errors at Week 12 were obtained from multiple imputation approach followed by robust regression model for handling of missing data. All available post-baseline data from Week 4 to Week 12 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: From Baseline to Week 12
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -31.7 (3.3) | -49.6 (3.3) | 1.3 (3.3)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Robust — Threshold for significance at 0.025 level for Bonferroni adjustment; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -32.9, 97.5% CI 2-sided [-43.4 to -22.5] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Robust — Threshold for significance at 0.025 level for Bonferroni adjustment; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -50.9, 97.5% CI 2-sided [-61.5 to -40.3] — Alirocumab 150 mg Q2W vs. Placebo

13. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 12- ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 12
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | 7.7 (1.8) | 9.9 (1.8) | 2.0 (1.8)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0241, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = 5.7, 97.5% CI 2-sided [0.0 to 11.3] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0022, Mixed Models Analysis — Threshold for significance at 0.025 level for Bonferroni adjustment; LS Mean Difference = 7.8, 97.5% CI 2-sided [2.1 to 13.5] — Alirocumab 150 mg Q2W vs. Placebo

14. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides (TGs) at Week 12: ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 12 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 12
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | -0.6 (3.7) | -18.0 (3.8) | -6.4 (3.7)
Statistical Analysis 1: Comparison: Alirocumab 150 mg Q4W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.2645, Regression, Robust — Threshold for significance at 0.025 level for Bonferroni adjustment; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = 5.9, 97.5% CI 2-sided [-5.9 to 17.7] — Alirocumab 150 mg Q4W vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 150 mg Q2W vs Placebo Q2W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0299, Regression, Robust — Threshold for significance at 0.025 level for Bonferroni adjustment; Adjusted Mean Difference = -11.6, 97.5% CI 2-sided [-23.5 to 0.4] — Alirocumab 150 mg Q2W vs. Placebo

15. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-1) at Week 12: ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 12
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment (Apo A-1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 150 mg Q4W | Alirocumab 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 54 | 53 | 56
percent change | 6.8 (1.6) | 9.1 (1.7) | 2.9 (1.6)

16. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 20, 24, 36, 48 and 64 -OLTP Analysis
Time Frame: Baseline, Weeks 20, 24, 36, 48 and 64
Population: Open-label treatment (OLT) population included all randomized participants who received at least one dose or part of dose of open-label investigational medicinal product. Here, "number analyzed" signifies participants with available data at each specified time-point.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Alirocumab 150mgQ4W/Up Q2W(After Alirocumab 150mgQ4W in DBTP): Participants who received alirocumab 150 mg Q4W during DBTP and completed DBTP, entered in OLTP and received alirocumab 150 mg Q4W from Week 12 up to Week 64. Alirocumab dose up-titrated to 150 mg Q2W at Week 24 (Week 12 of OLTP), when LDL-C levels ≥100 mg/dL (2.59 mmol/L) or ≥120 mg/dL (3.10 mmol/L) at Week 20 according to JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
- Alirocumab 150mgQ4W/Up Q2W(After Alirocumab 150mgQ2W in DBTP): Participants who received alirocumab 150 mg Q2W during DBTP and completed DBTP, entered in OLTP and received alirocumab 150 mg Q4W from Week 12 up to Week 64. Alirocumab dose up-titrated to 150 mg Q2W at Week 24 (Week 12 of OLTP), when LDL-C levels ≥100 mg/dL (2.59 mmol/L) or ≥120 mg/dL (3.10 mmol/L) at Week 20 according to JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
- Alirocumab 150mg Q4W/Up Q2W (After Placebo Q2W in DBTP): Participants who received Placebo Q2W during DBTP and completed DBTP, entered in OLTP and received alirocumab 150 mg Q4W from Week 12 up to Week 64. Alirocumab dose up-titrated to 150 mg Q2W at Week 24 (Week 12 of OLTP), when LDL-C levels ≥100 mg/dL (2.59 mmol/L) or ≥120 mg/dL (3.10 mmol/L) at Week 20 according to JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
Arm/Group | Alirocumab 150mgQ4W/Up Q2W(After Alirocumab 150mgQ4W in DBTP) | Alirocumab 150mgQ4W/Up Q2W(After Alirocumab 150mgQ2W in DBTP) | Alirocumab 150mg Q4W/Up Q2W (After Placebo Q2W in DBTP)
Number analyzed (Participants) | 54 | 50 | 54
Percent change
  Week 20: number analyzed (Participants) | 53 | 50 | 53
  Week 20 | -42.1 (20.1) | -47.8 (24.2) | -45.5 (20.5)
  Week 24: number analyzed (Participants) | 53 | 49 | 51
  Week 24 | -39.7 (20.4) | -46.0 (20.0) | -47.8 (21.7)
  Week 36: number analyzed (Participants) | 52 | 49 | 51
  Week 36 | -49.2 (19.4) | -51.5 (19.6) | -56.2 (18.8)
  Week 48: number analyzed (Participants) | 52 | 48 | 48
  Week 48 | -48.6 (21.6) | -53.9 (17.6) | -57.8 (17.4)
  Week 64: number analyzed (Participants) | 51 | 48 | 47
  Week 64 | -44.3 (22.8) | -55.2 (17.5) | -58.1 (19.6)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the end of study (up to Week 64) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are TEAEs that is AEs that developed/ worsened and death that occurred during 'treatment-emergent period' (time from first dose of study drug up to last dose of study drug +70 days). Analysis performed on safety population which included randomized participants who actually received at least 1 dose or partial dose of double-blind IMP injection for double-blind treatment period and at least 1 dose or partial dose of open-label IMP injection for open-label treatment period.
Groups:
- Double-blind Treatment Period: Placebo Q2W: Participants received Placebo (for alirocumab) SC injection Q2W added to lowest-strength statin therapy (atorvastatin 5 mg), stable non-statin LMT or diet therapy alone for 12 weeks.
- Double-blind Treatment Period: Alirocumab 150 mg Q4W: Participants received Alirocumab 150 mg SC injection Q4W alternating with placebo (for alirocumab) Q4W added to lowest-strength of statin therapy (atorvastatin 5 mg daily) stable non-statin LMT or diet therapy alone for 12 weeks.
- Double-blind Treatment Period: Alirocumab 150 mg Q2W: Participants received Alirocumab 150 mg SC injection Q2W added to lowest-strength statin therapy (atorvastatin 5 mg), stable non-statin LMT or diet therapy alone for 12 weeks.
- Open-label Treatment Period: Alirocumab 150 mg Q4W/Up Q2W: All participants received alirocumab 150 mg Q4W from the start of the open-label treatment period. Alirocumab dose up-titrated from 150 mg Q4W to 150 mg Q2W at Week 24 (Week 12 of OLTP), when LDL-C levels ≥ 100 mg/dL (2.59 mmol/L) or ≥ 120 mg/dL (3.10 mmol/L) at Week 20 according to JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
Arm/Group | Double-blind Treatment Period: Placebo Q2W | Double-blind Treatment Period: Alirocumab 150 mg Q4W | Double-blind Treatment Period: Alirocumab 150 mg Q2W | Open-label Treatment Period: Alirocumab 150 mg Q4W/Up Q2W
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/54 | 1/53 | 0/158
Serious Adverse Events (participants affected / at risk) | 1/56 | 1/54 | 2/53 | 12/158
Other Adverse Events (participants affected / at risk) | 14/56 | 11/54 | 13/53 | 72/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Period: Placebo Q2W (N=56) | Double-blind Treatment Period: Alirocumab 150 mg Q4W (N=54) | Double-blind Treatment Period: Alirocumab 150 mg Q2W (N=53) | Open-label Treatment Period: Alirocumab 150 mg Q4W/Up Q2W (N=158)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Facial spasm (Nervous system disorders) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Period: Placebo Q2W (N=56) | Double-blind Treatment Period: Alirocumab 150 mg Q4W (N=54) | Double-blind Treatment Period: Alirocumab 150 mg Q2W (N=53) | Open-label Treatment Period: Alirocumab 150 mg Q4W/Up Q2W (N=158)
Pharyngitis (Infections and infestations) | 0 | 3 | 0 | 5
Viral upper respiratory tract infection (Infections and infestations) | 9 | 8 | 8 | 54
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 8
Non-cardiac chest pain (General disorders) | 1 | 0 | 4 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT02584504/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT02584504/SAP_001.pdf